CLINICAL TRIAL: NCT06112301
Title: Pivotal, Clinical Study for the Accuracy Evaluation of the IdentiClone Dx IGH Assay
Status: Completed | Type: Observational
Sponsor: Invivoscribe, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVS-108-001
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: B-Cell Lymphoproliferative Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Deidentified residual DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- B-Cell Positive Lymphoproliferative Disorders: DNA Samples for subjects with B-Cell Positive Lymphoproliferative Disorders
  Interventions: Diagnostic Test: IdentiClone Dx IGH (IC IGH Dx) Assay
- B-Cell Negative Lymphoproliferative Disorders: DNA Samples for subjects suspected of B-Cell Positive Lymphoproliferative Disorders with negative B-Cell Clonality testing
  Interventions: Diagnostic Test: IdentiClone Dx IGH (IC IGH Dx) Assay

INTERVENTIONS:
Diagnostic Test: IdentiClone Dx IGH (IC IGH Dx) Assay — The IdentiClone Dx IGH Assay is an in vitro diagnostic product intended for qualitative, capillary electrophoresis based-detection of clonality in immunoglobulin heavy chain gene rearrangements (IGH) in peripheral blood specimens as an adjunctive method for the diagnosis of B-cell lymphoproliferative disease

SUMMARY:
This protocol describes the pivotal accuracy study for the IdentiClone Dx IGH (IC IGH Dx) Assay. The intent of the accuracy study is to demonstrate agreement between the results of the IC IGH Dx Assay and a predicate devise or assay on retrospective and residual de-identified DNA extracted from peripheral blood (PB) samples from individuals with suspected B-Cell Lymphoproliferations. The predicate device will be the LymphoTrack Dx IGH (FR1/FR2/FR3) Assays - MiSeq (LT Dx IGH-CE-IVD), which is a CE-IVD assay with a similar intended use as the IC IGH Assay on the same sample type.

ELIGIBILITY:
Inclusion Criteria:

1. DNA extracted from Peripheral Blood (PB) with EDTA as anticoagulant with minimum total DNA ≥ 2 µg with concentration at ≥ 50ng/µl
2. DNA extracted from PB specimens no more than 7 days
3. DNA stored at -15°C to -30°C up to 5 years
4. Donor Age: ≥ 18
5. For positive sample, DNA from PB of subjects diagnosed (at the time the specimen was drawn) with Lymphoproliferative disease, with:

   1. ICD 10 Codes: C8300, C8330, C8510 or other B-cell leukemia/lymphoma diagnosis
   2. B-cell Lymphoproliferative disease diagnosis per collection site procedure (i.e. SNOMED)
6. For negative sample, DNA from PB of subjects suspected of Lymphoproliferative disease

Exclusion Criteria:

1. PB specimens that have been frozen prior to extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from subjects with diagnosed B-Cell Lymphoproliferative disorders or suspected of B-Cell Lymphoproliferative disorders with negative B-Cell Clonality Testing results
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
% Agreement | Through Study Completion at one year
  Agreement between the results of the Invivoscribe IdentiClone Dx IGH Assay and the LymphoTrack Dx IGH (FR1/FR2/FR3) Assays - MiSeq by assessing the positive and negative percent agreement between the two assays.

CONTACTS AND LOCATIONS:
Locations (3):
- Invivoscribe, Inc., San Diego, California, United States
- LabPMM GmbH, Hallbergmoos, Germany
- LabPMM GK, Kawasaki-shi, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No